CLINICAL TRIAL: NCT01056016
Title: Disseminating a Model Intervention to Promote Improved ADHD Care in the Community
Brief Title: Disseminating a Model Intervention to Promote Improved Attention-deficit Hyperactivity Disorder (ADHD) Care in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Jeff Epstein, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R21MH082714 (NIH)
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait-list control (No Intervention): Wait-list control group
- ADHD Collaborative Intervention (Experimental): This intervention includes mapping and redesign of office flow to facilitate adherence to AAP ADHD guidelines as well as didactic sessions related to diagnosis and treatment of ADHD. Didactics emphasize the importance of obtaining parent and teacher behavioral ratings (e.g. Vanderbilt ADHD Rating Scales) at the time of the initial assessment for ADHD and during follow-up after initiating medication treatment and making a Diagnostic and Statistical Manual-IV (DSM-IV) based ADHD diagnosis. Practices are given a web-based ADHD portal to assist them in creating a patient registry and to help in obtaining parent and teacher ratings scales. The intervention lasts for 6 months.
  Interventions: Other: ADHD Collaborative

INTERVENTIONS:
Other: ADHD Collaborative — This intervention includes mapping and redesign of office flow to facilitate adherence to AAP ADHD guidelines as well as didactic sessions related to diagnosis and treatment of ADHD. Didactics emphasize the importance of obtaining parent and teacher behavioral ratings (e.g. Vanderbilt ADHD Rating Scales) at the time of the initial assessment for ADHD and during follow-up after initiating medication treatment and making a DSM-IV based ADHD diagnosis. Practices are given a web-based ADHD portal to assist them in creating a patient registry and to help in obtaining parent and teacher ratings scales.
  Arms: ADHD Collaborative Intervention

SUMMARY:
The American Academy of Pediatrics (AAP) has established a set of consensus guidelines for pediatricians to follow. These guidelines can be challenging to implement in typical community-based practices. Cincinnati Children's Hospital Medical Center (CCHMC) has developed a program called the ADHD Collaborative to promote the adoption of these guidelines among community pediatricians. The program focuses on modifying the office system using academic detailing and quality improvement (QI) methodology to accommodate prescribed practice changes. The ADHD Collaborative has been very successful at recruiting practices in the Greater Cincinnati area, changing practice behaviors, and sustaining these practice behaviors over time at minimal cost to the project and to the office practice. Now that sustainability and effectiveness have been established, the next step is to modify the ADHD Collaborative model to make it amenable to widespread dissemination. The primary goal of the proposed study is to modify the ADHD Collaborative intervention to make it transportable and then evaluate this version in terms of effectiveness, consumer satisfaction, and costs.. A transportable intervention is described that utilizes telehealth videoconferencing, a web portal, and long-distance data collection. Initially, three pediatric practices will be recruited to test and refine the distal intervention delivery methodology. Then, eight new pediatric practices will be randomly assigned to receive the distal intervention or to a control group (treatment as usual). Information about pediatric practice behavior will be collected at baseline, 6-months, and 1-year post-baseline. The study design will allow for a preliminary assessment of the feasibility and effectiveness of the distal intervention in terms of rates of evidence-based practice behaviors to patients, change in pediatrician attitudes, consumer satisfaction, and costs.

ELIGIBILITY:
Inclusion Criteria:

* pediatric practice with at least 2 physicians

Exclusion Criteria:

* no electronic billing system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Epstein JN, Langberg JM, Lichtenstein PK, Mainwaring BA, Luzader CP, Stark LJ. Community-wide intervention to improve the attention-deficit/hyperactivity disorder assessment and treatment practices of community physicians. Pediatrics. 2008 Jul;122(1):19-27. doi: 10.1542/peds.2007-2704. PMID 18595982
- [Result] Epstein JN, Langberg JM, Lichtenstein PK, Kolb R, Altaye M, Simon JO. Use of an Internet portal to improve community-based pediatric ADHD care: a cluster randomized trial. Pediatrics. 2011 Nov;128(5):e1201-8. doi: 10.1542/peds.2011-0872. Epub 2011 Oct 17. PMID 22007005

RESULTS

PARTICIPANT FLOW:
Groups:
- ADHD Collaborative Intervention: This intervention includes mapping and redesign of office flow to facilitate adherence to American Academy of Pediatrics (AAP) ADHD guidelines as well as didactic sessions related to diagnosis and treatment of ADHD. Didactics include the importance of obtaining parent and teacher behavioral ratings at the time of the initial assessment for ADHD and during follow-up after initiating medication treatment and making a DSM-IV based ADHD diagnosis. Practices are given a web-based ADHD portal to assist them in creating a patient registry and to help in obtaining parent and teacher ratings scales. The intervention lasts for 6 months.
  ADHD Collaborative: This intervention includes mapping and redesign of office flow to facilitate adherence to AAP ADHD guidelines as well as didactic sessions related to diagnosis and treatment of ADHD. Didactics emphasize the importance of obtaining parent and teacher behavioral ratings (e.g. Vanderbilt ADHD Rating Scales) at the time of the initial
Period: Overall Study
Arm/Group | Wait-list Control | ADHD Collaborative Intervention
Started | 22 (22 pediatricians were at 4 practices; practices were unit of randomization) | 27 (27 pediatricians were at 4 practices; practices were unit of randomization)
Completed | 20 | 26
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- ADHD Collaborative Intervention: This intervention includes mapping and redesign of office flow to facilitate adherence to AAP ADHD guidelines as well as didactic sessions related to diagnosis and treatment of ADHD. Didactics emphasize the importance of obtaining parent and teacher behavioral ratings (e.g. Vanderbilt ADHD Rating Scales) at the time of the initial assessment for ADHD and during follow-up after initiating medication treatment and making a DSM-IV based ADHD diagnosis. Practices are given a web-based ADHD portal to assist them in creating a patient registry and to help in obtaining parent and teacher ratings scales. The intervention lasts for 6 months.
  ADHD Collaborative: This intervention includes mapping and redesign of office flow to facilitate adherence to AAP ADHD guidelines as well as didactic sessions related to diagnosis and treatment of ADHD. Didactics emphasize the importance of obtaining parent and teacher behavioral ratings (e.g. Vanderbilt ADHD Rating Scales) at the time of the initial
- Total: Total of all reporting groups
Arm/Group | Wait-list Control | ADHD Collaborative Intervention | Total
Number analyzed (Participants) | 22 | 27 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.0 (10.3) | 46.6 (11.3) | 46.8 (10.7)
Gender [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 7 | 13 | 20
Region of Enrollment [Number; unit: participants]
  United States | 22 | 27 | 49

OUTCOME MEASURES:

1. Primary Outcome: Physician ADHD Practice Behavior
Description: Percentage of patients across pediatricians in each randomized group for whom the pediatrician collected teacher ratings to monitor treatment response
Time Frame: Baseline and 6 months
Population: Patient chart reviews were conducted with 174 patients in the ADHD Collaborative Intervention group and 64 patients in the Wait-list control group
Measure: Mean (Standard Deviation); unit: percentage of patients
Arm/Group | Wait-list Control | ADHD Collaborative Intervention
Number analyzed (Participants) | 22 | 27
percentage of patients
  Baseline | 0 (0) | 0 (0)
  6-months | 6.3 (25.0) | 38.7 (36.1)
Statistical Analysis 1: Comparison: Wait-list Control vs ADHD Collaborative Intervention; The percentage of patients with whom pediatrician in each group utilized each practice behavior at baseline and 6-months was computed. The reported statistical analysis did not account potential clustering due to the small number of practices in this study; Test type: Superiority or Other; p = .003, t-test, 2 sided; Mean Difference (Net) = 32.4

ADVERSE EVENTS:
Description: Participants in each Arm/Group were not monitored for adverse events.
Arm/Group | Wait-list Control | ADHD Collaborative Intervention
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No